CLINICAL TRIAL: NCT05079789
Title: Randomized, Controlled Interventional Trial to Investigate the Efficacy of Amiloride for the Treatment of Edema in Human Nephrotic Syndrome
Brief Title: Amiloride in Nephrotic Syndrome
Acronym: AMILOR
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Low recruiting rate and decision to evaluate as pilot study
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, Dr. Anja Schork, Clinincal Investigator, Project management, University Hospital Tuebingen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AmiloridNS-01; 2019-002607-18 (EudraCT Number)
Record Dates: First submitted 2021-10-02; First posted 2021-10-15 (Actual); Results first posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Nephrotic Syndrome; Edema; Sodium Retention
Keywords: Nephrotic Syndrome; ENaC; Diuretic therapy; Amiloride; Proteasuria
MeSH Terms: conditions — Nephrotic Syndrome; Edema; Hypernatremia | interventions — Amiloride; Furosemide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Amiloride (Experimental): Treatment wirh Amiloride, start dose 5 mg
  Interventions: Drug: Amiloride
- Furosemide (Active Comparator): Treatment with Furosemide, start dose 40 mg
  Interventions: Drug: Furosemide

INTERVENTIONS:
Drug: Amiloride — Treatment with amiloride, start dose 5 mg
  Arms: Amiloride
Drug: Furosemide — Treatment with furosemide, start dose 40 mg
  Arms: Furosemide

SUMMARY:
The AMILOR study compares treatment of edema in nephrotic syndrome with Amiloride vs. Furosemide.

DETAILED DESCRIPTION:
The monocenter randomized-controlled AMILOR trial investigates the efficacy of the ENaC blocker amiloride in reducing edema in nephrotic syndrome compared with standard therapy with the loop diuretic furosemide.

Patients with acute nephrotic syndrome are randomized to receive amiloride (starting dose 5 mg) or furosemide (starting dose 40 mg) for 16 days. The target number of patients is n = 18 per arm. Exclusion criteria include GFR <30ml/min/1.73m², AKIN 1 and 2, hypotension, hyper-/ hypokalemia, and hyponatremia. Overhydration is quantified by bioimpedance spectroscopy. Depending on the course of overhydration, dose adjustments (day 2, 5, 8, 12) or addition of HCT (day 8) are performed during the course of the study.

Primary endpoint is decrease in overhydration at day 8, secondary endpoints include decrease in overhydration at day 16, as well as body weight, edema volume, blood pressure, urine volume, natriuresis at day 8 and 16, and need for dose adjustments and co-medication with HCT. Plasma potassium, sodium, and creatinine concentrations are measured as safety parameters.

ELIGIBILITY:
Inclusion Criteria:

1. Acute nephrotic syndrome with proteinuria > 3 g/day and formation of edema.
2. Age ≥ 18 years at the time of signing the informed consent.
3. Understand and voluntarily sign an informed consent document prior to any study related assessments/procedures.
4. Ability to adhere to the study visit schedule and other protocol requirements.
5. Use of adequate thrombosis prophylaxis due to the increased risk of thrombosis in nephrotic syndrome and the expected fluctuations in volume balance during study participation.
6. Subject (male or female) is willing to use highly effective methods of contraception according to the "Clinical trial fertility group" recommendations.
7. Female Patients of childbearing potential (WOCBP) must agree to pregnancy testing before inclusion in the study.
8. Female Patients must agree to abstain from breastfeeding during study participation and 28 days after study drug discontinuation.
9. All subjects must agree not to share medication.

Exclusion Criteria:

1. Severe reduction of kidney function: Creatinine clearance or calculated GFR < 30 mL/min/1.73m² or acute kidney injury KDIGO stage 2 or 3 or anuria.
2. Hypovolemia or dehydration.
3. Uncontrolled diabetes mellitus.
4. Hypotension, systolic blood pressure < 90 mmHg.
5. Hyperkalemia, plasma potassium concentration > 4.8 mmol/l.
6. Hypokalemia, plasma potassium concentration < 3.3 mmol/l.
7. Hyponatremia, plasma sodium concentration < 128 mmol/l.
8. Hypercalcemia, ionized calcium > 2.0 mmol/l or total albumin corrected calcium > 3.0 mmol/l.
9. Signs of cardiac decompensation (orthopnoe, dyspnoe NYHA IV).
10. Hepatic coma or precoma.
11. Symptoms of gout.
12. Current therapy with potassium-sparing diuretics (e.g. spironolactone) or potassium supplements.
13. Women during pregnancy and lactation.
14. History of hypersensitivity to the investigational medicinal product, comparator or co-medication or to any drug with similar chemical structure or to any excipient present in the pharmaceutical form of the investigational medicinal product, comparator or co-medication.
15. Any other clinical condition that would jeopardize the patient's safety while participating in this clinical trial.
16. Active participation in other clinical trials or observation period of competing trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-06-08 (Actual); Primary Completion 2022-11-05 (Actual); Study Completion 2022-11-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ferruh Artunc, Prof., MD, Principal Investigator — University Hospital Tuebingen
Locations (1):
- University Hospital Tuebingen, Tübingen, Baden-Wurttemberg, Germany

REFERENCES:
- [Background] Artunc F, Worn M, Schork A, Bohnert BN. Proteasuria-The impact of active urinary proteases on sodium retention in nephrotic syndrome. Acta Physiol (Oxf). 2019 Apr;225(4):e13249. doi: 10.1111/apha.13249. Epub 2019 Jan 18. PMID 30597733
- See also: Homepage working group Prof. Artunc — https://www.medizin.uni-tuebingen.de/de/das-klinikum/einrichtungen/kliniken/medizinische-klinik/innere-medizin-iv/forschung/nierenphysiologie

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Amiloride | Furosemide
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Amiloride | Furosemide | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 8 | 16
  >=65 years | 2 | 2 | 4
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 51 [46 to 53] | 50 [25 to 58] | 51 [36 to 55]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 7
  Male | 5 | 8 | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: European | 9 | 10 | 19
  Ethnicity: Indian | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Germany | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Decrease of Overhydration, %ECW After 8 Days
Description: Decrease of overhydration (OH) measured by bioimpedance spectroscopy, expressed as percent of extracellular water (%ECW)
Time Frame: 8 days
Measure: Median (Inter-Quartile Range); unit: %ECW
Arm/Group | Amiloride | Furosemide
Number analyzed (Participants) | 10 | 10
%ECW | 1.95 [0.80 to 6.40] | 5.15 [0.90 to 8.30]

2. Secondary Outcome: Decrease of Overhydration, %ECW After 16 Days
Description: as for outcome 1
Time Frame: 16 days
Measure: Median (Inter-Quartile Range); unit: %ECW
Arm/Group | Amiloride | Furosemide
Number analyzed (Participants) | 9 | 10
%ECW | 10.10 [1.30 to 14.40] | 7.40 [2.80 to 10.10]

3. Secondary Outcome: Decrease of Body Weight, kg
Description: Decrease of body weight after 8 days
Time Frame: 8 days
Measure: Median (Inter-Quartile Range); unit: kg
Arm/Group | Amiloride | Furosemide
Number analyzed (Participants) | 10 | 10
kg | 3.8 [1.7 to 7.2] | 2.0 [1.5 to 4.6]

ADVERSE EVENTS:
Time Frame: 23 days for everey subject
Arm/Group | Amiloride | Furosemide
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 1/10 | 4/10
Other Adverse Events (participants affected / at risk) | 9/10 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Amiloride (N=10) | Furosemide (N=10)
delayed discharge from hospital due to macrohematuria after kidneybiopsy (Surgical and medical procedures) | 1 (1) | 0 (0) — delayed discharge from hospital due to macrohematuria after kidney biopsy
myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) — myocardial infarction
pericardial effusion with in-hospital monitoring (Cardiac disorders) | 0 (0) | 1 (1) — pericardial effusion with in-hospital monitoring
abdominal pain with diarrhea with inhospital treatment (Gastrointestinal disorders) | 0 (0) | 1 (1) — abdominal pain with diarrhea with inhospital treatment
AKI stage 2 with in-hospital treatment (Renal and urinary disorders) | 0 (0) | 1 (1) — AKI stage 2 with in-hospital treatment
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Amiloride (N=10) | Furosemide (N=10)
planned hospitalization for kidney biopsy (Surgical and medical procedures) | 2 (2) | 3 (3) — planned hospitalization for kidney biopsy
dizziness (Nervous system disorders) | 0 (0) | 1 (1) — dizziness
headache (Nervous system disorders) | 0 (0) | 1 (1) — headache
nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) — nausea
epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) — epistaxis
elevated liver enzymes (Hepatobiliary disorders) | 0 (0) | 1 (1) — elevated liver enzymes
rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — rash
urinary infection (Renal and urinary disorders) | 1 (1) | 0 (0) — urinary infection
hypervolemia (worsening) (Renal and urinary disorders) | 1 (1) | 0 (0) — hypervolemia (worsening)
SARS CoV 2 infection (Infections and infestations) | 2 (2) | 1 (1) — SARS CoV 2 infection
cramps of legs and hands (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — cramps of legs and hands

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2021-03-01): https://cdn.clinicaltrials.gov/large-docs/89/NCT05079789/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-17): https://cdn.clinicaltrials.gov/large-docs/89/NCT05079789/SAP_001.pdf